CLINICAL TRIAL: NCT06722131
Title: Création d'Une biothèque de prélèvements de Patients présentant Une Pathologie Infectieuse
Brief Title: Biobank of Samples From Patients With Infectious Diseases
Acronym: INFECTIOTEK
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240413
Record Dates: First submitted 2024-12-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Infectious Diseases
Keywords: Biobank; Bacterial, viral and fungal diseases
MeSH Terms: conditions — Communicable Diseases; Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling
  In addition, infection site sampling according to pathology :
  * Urine
  * Stool
  * cerebrospinal fluid
  * Sputum or bronchoalveolar lavage liquid
  * Nasopharyngeal swab
  * Genital swab
  * Skin swab
  * Biopsy (a fragment of a lung, kidney or brain biopsy if performed)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with an infectious disease
  Interventions: Other: Sampling

INTERVENTIONS:
Other: Sampling — Additional biological sampling at the same time as routine-care samples taken in the context of the diagnosis of the infectious disease and if planned at one and 12 months of follow-up
  * The considered samples are as follows :
    * Blood sample tubes (5 x 5 mL tubes, i.e. 25 mL)
    * Infection site sample if applicable :
  * Urine (10 mL)
  * Stool (1 mL)
  * CSF (1 mL)
  * Sputum (1 mL) or bronchoalveolar lavage fluid (10 mL)
  * Nasopharyngeal swab (one swab)
  * Genital swab (one swab)
  * Skin swab (one swab)
  * Biopsy (a fragment of a lung, kidney or brain biopsy, if performed)

SUMMARY:
The aim of the INFECTIOTEK biobank will be to prospectively build a biobank of multiple biological samples from patients with infectious diseases in order to identify diagnostic and prognostic biomarkers, genetic susceptibility factors and immune response mechanisms in such diseases.

The population of the study will consist of patients treated in the Infectious Diseases Departments of Saint-Louis and Lariboisière Hospitals, with a diagnosis of infectious disease, and who have biological samples in the context of their routine medical care.

The diseases studied in this research project are bacterial infections (urinary tract infections, neurologic infections, sexually transmitted infections, pulmonary infections), viral infections (HIV, hepatitis, respiratory viruses, viruses affecting immunocompromised patients) and fungal infections (Aspergillus, Mucorales, Cryptococcus). These diseases are the domains of expertise and research of the clinical and biological teams at the Saint-Louis and Lariboisière hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Diagnosed with one of the following infectious diseases :

  * Infection with HIV-1 or HIV-2, or person at risk of infection with HIV
  * Viral hepatitis (HAV, HBV, HCV, HDV, HEV)
  * Pulmonary infections: bacterial (notably Nocardia), viral (Influenza, RSV, SARS-CoV-2, Adenovirus), fungal (Aspergillus, Mucorales)
  * Urinary tract infections
  * Sexually transmitted infections (Neisseria gonorrheae, Chlamydia trachomatis, Mycoplasma genitalium, Treponema pallidum)
  * Neuromeningeal infections: (Neisseria meningitidis, Streptococcus pneumoniae), viral (HSV, VZV), fungal (Cryptococcus).
  * Infections affecting immunocompromised patients: herpes viruses (HSV, VZV, CMV, EBV), polyomavirus BK
  * Emerging pathogen X (in the event of an epidemic)
  * Signature of research consent form
  * Health coverage with social security system or state medical aid

Exclusion Criteria:

* Refusal to participate
* Inability to give consent (cognitive impairment etc...)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated in the Infectious Diseases Departments of Saint-Louis and Lariboisière Hospitals, with a diagnosis of infectious disease, and who have biological samples in the context of their routine medical care
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performances of new biomarkers to identify infection | At diagnosis
  Sensitivity, Specificity, Positive Predictive Value, Negative Predictive Value, Positive Likelihood Ratio, Negative Likelihood Ratio of the new biomarker

SECONDARY OUTCOMES:
Description of pathophysiological phenomena | Until 12 months
  Resistance mechanisms, virulence parameters, immune responses to the infectious agent, susceptibility factors to infections
Description of prognostic biomarkers | Until 12 months